CLINICAL TRIAL: NCT07180290
Title: Evaluation of the ChronoS Therapy on the Severity of Sleep Disturbances Among Patients With Mood Disorders: A Within-subjects Study
Acronym: CRHONOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D22_EPI0028
Record Dates: First submitted 2025-01-31; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Insomnia Due to Mental Disorder
Keywords: Insomnia; Mood disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mood Disorders | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bipolar disorder (Experimental): Bipolar disorder is defined by the DSM-5 as the experience of episodes of depression or anhedonia (i.e., a lack of interest or pleasure in activities) and at least four additional symptoms: decreased energy; psychomotor slowing or psychomotor restlessness; changes in appetite and weight; sleep disturbance (from insomnia to hypersomnia); difficulty concentrating and/or inability to make everyday decisions; feelings of worthlessness and/or excessive guilt; and suicidal ideation and attempts.
  Interventions: Behavioral: Psychotherapy
- Unipolar disorder (Experimental): Unipolar disorder is defined by the DSM-5 as the experience of 5 or more of the following symptoms, at least once per day, and for a period that's longer than 2 weeks:
  * Sadness or irritability, lasting most of the day
  * Loss of interest in the majority of activities that were enjoyable before
  * Change in appetite, or sudden weight loss/gain
  * Difficulty falling asleep, or wanting to sleep more than before
  * Feelings of restlessness
  * Lack of energy and increased tiredness
  * Feelings of worthlessness or guilt, often linking to things that normally wouldn't have this kind of effect
  * Difficulty concentrating, making decisions and thinking
  * Suicidal or self-harming thoughts
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Session 1 : Introduction and awareness of the sleep-wake link Session 2 : Awareness of day/night habits and behaviors Session 3 : Awareness of sleep/wake rhythms and sleepiness signals Session 4 : Awareness of the night/bed/sleep association Session 5 : Awareness of emotions and thoughts related to sleep Session 6 : Awareness of possible alternatives Session 7 : Awareness of one's relationship to sleep Session 8 : Awareness of future benefits

SUMMARY:
A new psychotherapy has been developed within the Psychiatry, Sleep and Chronobiology Reference Center (ChronoS) since January 2022.Results have shown relevant clinical interest on insomnia symptoms, as well on mood, anxiety and hypervigilance, according to the observation of the center's team (nurses, psychologists, psychiatrists and somnologist) In order to evaluate the effectiveness of this psychotherapy, the investigators would like to carry a multimodal approach on the severity of insomnia in patients with mood disorders.

DETAILED DESCRIPTION:
Insomnia affects 85% of patients with a mood disorder during depressive phases and more than 50% will suffer from insomnia symptoms after remission. The treatment of insomnia with mood disorders represents a major therapeutic issue.European recommendations suggest that cognitive behavioural therapy for insomnia (iCBT) as the first-line reference treatment for chronic insomnia disorder.

However, only 38% of patients respond positively to the treatment at 24 months, while 50% of patients with insomnia disorder and mood disorder do not respond to the treatment.

The two main reasons are reported :

1) insomnia often hide circadian disruption, or 2) patients often-present states of emotional dysregulation known as hyperarousal or hyperarousal, which result in a partial response to treatment.

A new psychotherapy was developed within the Psychiatry, Sleep and Chronobiology Reference Center (ChronoS) integrating:

1. Interpersonal and Social Rhythm Therapy
2. Chronotherapies to regulate sleep/wake cycles
3. Positive mental imagery for stress management
4. Mindfulness therapy for both stress and hyperarousal state management

iCBT is also adapted to a certain extent to sleep restriction to avoid sleep deprivation which is strongly linked to relapse in bipolar disorders.

This psychotherapy is being practiced within the Psychiatry, Sleep and Chronobiology Reference Center (ChronoS) since January 2022, and results have shown relevant clinical interest on insomnia symptoms, as well as on mood, anxiety and hypervigilance, according to the observation of the team center (nurses, psychologists, psychiatrists and somnologist) Thus, the investigators wish to carry out a before/after study to evaluate the effectiveness of this psychotherapy with multimodal approaches on the severity of insomnia in patients with mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old
* Diagnosed with

  1. A mood disorder (bipolar or unipolar) recognized in the DSM-5
  2. Chronic insomnia disorder recognized in the DSM-5
* Must have obtained a score ≥ 8 on the ISI scale evaluated by the clinician, that indicates at least an insomnia of mild intensity

Exclusion Criteria :

* Patients aged under 18 years old
* Patients with psychotic disorder
* Patients who have previously undergone CBT insomnia or other targeted cognitive behavioral therapy
* Patients under guardianship, curatorship or protection of the court

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  brief self report questionnaire to assess the severity of insomnia cases

SECONDARY OUTCOMES:
Seasonal Pattern Assessment Questionnaire (SPAQ) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  questionnaire to evaluate seasonal effects on mood and behavior
Morningness-Eveningness Questionnaire (MEQ) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  Scale used to evaluate chronotype
The Berlin Questionnaire | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  Questionnaire used to assess the risk of developing sleep apnea syndrome.
Pittsburgh Sleep Quality Index | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  self-report instrument used to evaluate posttraumatic stress disorder (PTSD)
The Epworth Sleepiness Scale (ESS) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  self-administered questionnaire used by doctors to assess daytime sleepiness
The Disturbing Dream and Nightmare Severity Index (DDNSI) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  self-retrospective measure of current nightmare and disturbing dream frequency and severity
Wakefulness after sleep onset (WASO) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  measurement used to assess a person's sleep
A sleep fragmentation index (SFI) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  calculate the total number of awakenings/shifts divided by the total sleep time in hours
Sleep efficiency (SE) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  Ratio of total sleep time (TST) to time in bed (TIB), duration divided by the bed duration
Hyperarousal Scale (HAS) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  self-report of symptoms initially described in insomnia patients
The Hospital Anxiety and Depression Scale (HADS) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  Scale used to assess anxiety and depression symptoms in patients
Quick Inventory of Depressive Symptomatology (QIDS) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  brief self report tool used to evaluation the symptoms of depression
Generalized Anxiety Disorder 7 (GAD-7) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  self-reported questionnaire for screening and severity measuring of generalized anxiety disorder
The Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  A 7 point scale used to measure severity of depression in individuals 18 years and older. Each item is rated on a 7-point scale
Multidimensional Assessment of Thymic States) (MATHYS) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  scale used to define mood states dimensionally
Young Mania Rating Scale (YMRS) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  rating scales to assess manic symptoms
The Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  Scale used to quantify the severity of suicidal ideation and behavior
Consumption of self medicated sleeping pills | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  type,dosage, frequency of consumption of sleeping pills
Psychotropic treatment | Baseline visit : at participants' inclusion Visit 1: alongside 1st session of the therapy Visit 2: after the 4th session of the therapy Visit 3: after the last session (8th) of the therapy Visit 4 : 3 months after the end of the therapy
  frequency and impact of psychotropic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexis GEOFFROY, Professor of psychiatry, Study Director — GHU Paris Psychiatrie et Neurosciences
Locations (1):
- Centre CHRONOS, Paris, France